CLINICAL TRIAL: NCT01576328
Title: A Randomized, Placebo-Controlled Dose-Escalation Study to Assess the Safety and Tolerability of a Single Intravenous Infusion of Allogeneic Mesenchymal Precursor Cells (MPCs) in Patients With Type 2 Diabetes Sub-optimally Controlled on Metformin
Brief Title: Safety Study of Mesenchymal Precursor Cells in Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSB-DM003
Record Dates: First submitted 2012-04-09; First posted 2012-04-12 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): MPC dose 1 or Placebo
  Interventions: Drug: Mesenchymal Precursor Cells (MPCs)
- Cohort 2 (Experimental): MPC dose 2 or Placebo
  Interventions: Drug: Mesenchymal Precursor Cells (MPCs)
- Cohort 3 (Experimental): MPC dose 3 or Placebo
  Interventions: Drug: Mesenchymal Precursor Cells (MPCs)

INTERVENTIONS:
Drug: Mesenchymal Precursor Cells (MPCs) — Single intravenous infusion of MPCs Dose 1
  Arms: Cohort 1
Drug: Mesenchymal Precursor Cells (MPCs) — Single intravenous infusion of MPCs Dose 2
  Arms: Cohort 2
Drug: Mesenchymal Precursor Cells (MPCs) — Single intravenous infusion of MPCs Dose 3
  Arms: Cohort 3

SUMMARY:
This study is being conducted to assess the overall safety and tolerability of a single intravenous infusion of three doses of Mesenchymal Precursor Cells versus Placebo in subjects with Type 2 Diabetes inadequately controlled on Metformin.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female subjects who are ≥ 18 and ≤ 80 years old
* Subjects diagnosed with type 2 diabetes at least one year prior to Screening and receiving a stable, therapeutic dose of metformin > 1500 mg/day according to local prescribing information for at least 3 months prior to Screening or the highest tolerated dose > 1000 mg/day documented in the subject's history
* HbA1c > 7.0% and < 10.5% at Screening
* C-peptide > 0.8 ng/mL at Screening
* Body mass index (BMI) > 22 and < 45 kg/m2 at Screening
* Body weight < 150 kg at Screening

Key Exclusion Criteria:

* Prior participation in any stem cell study
* Women who are pregnant, intending to become pregnant during the study period or currently lactating
* History of active substance abuse (including alcohol) within the past 2 years. Current alcohol abuse is defined as daily consumption of >3 alcoholic beverage. Current cigarette smoking > 10 cigarettes per day
* Severe hypoglycemia (defined as requiring third party assistance) or repeated and/or frequent hypoglycemia episodes (> 2 episodes/week) within one month prior to Screening
* Patients receiving treatment for type 2 diabetes with diet and exercise alone, insulin therapy within 6 months of Screening except if used transiently for < 7 days for intercurrent illness or any other anti-diabetic medication except metformin within 3 months of Screening
* Any concurrent medical condition/disorder or clinically symptomatic cardiovascular, gastrointestinal (including pancreatitis), renal, hematological, pulmonary, acute or chronic infectious disease, active retinal disease, or other disorder which in the Investigator's opinion would interfere with the subject's ability to complete the trial, would require administration of treatment that could affect the interpretation of the safety and efficacy variables or would preclude safe involvement in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Primary objective of the study is to assess the safety and tolerability of MPC therapy | 116 Weeks
  Outcomes include the measurement of the following safety parameters:
  * Adverse events and serious adverse events(including hypoglycemia)
  * Vital signs (BP, HR, RR, O2 saturation)
  * Physical examinations
  * Results of clinical laboratory tests (hematology, biochemistry, and urinalysis, flow cytometry Class I and Class II PRA % with specificity, antibovine and antimurine antibody analysis)
  * Pulmonary function test
  * Electrocardiograms
  * Chest X-ray
  * Fundus oculi examination

CONTACTS AND LOCATIONS:
Overall Officials: K Segal, PhD, Study Director — Mesoblast, Ltd.
Locations (18):
- United States (18):
  - SC Clinical Research, Garden Grove, California
  - Diabetes Research Institute, Miami, Florida
  - Compass Research, Orlando, Florida
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Tulane University Medical Center, New Orleans, Louisiana
  - Big Sky Clinical Research, Butte, Montana
  - Desert Endocrinology Clinical Research Center-Henderson, Henderson, Nevada
  - Alliance Against Diabetes/AAD Clinical Research, Las Vegas, Nevada
  - Active Practices and Research, Newington, New Hampshire
  - The Carl and Edyth Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Providence Health Partners - Center for Clinical Reseach, Dayton, Ohio
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - West Houston Clinical Research Services, Houston, Texas
  - Paragon Research Center, San Antonio, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - National Clinical Research - Norfolk, Inc, Norfolk, Virginia
  - National Clinical Research - Richmond, Inc., Richmond, Virginia
  - Capital Clinical Research Center, Olympia, Washington

REFERENCES:
- [Derived] Skyler JS, Fonseca VA, Segal KR, Rosenstock J; MSB-DM003 Investigators. Allogeneic Mesenchymal Precursor Cells in Type 2 Diabetes: A Randomized, Placebo-Controlled, Dose-Escalation Safety and Tolerability Pilot Study. Diabetes Care. 2015 Sep;38(9):1742-9. doi: 10.2337/dc14-2830. Epub 2015 Jul 7. PMID 26153271